CLINICAL TRIAL: NCT06446115
Title: Decreasing Chemotherapy Induced Distress Using Immersive Virtual Reality in Patients With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE3124
Record Dates: First submitted 2024-05-29; First posted 2024-06-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Malignant Neoplasm; Cancer
Keywords: Virtual Reality; Chemotherapy
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: This is a two-arm, randomized 1:1, pilot study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): Participants will be asked to use a headset device during 15 to 30 minutes while receiving a chemotherapy infusion. Participants have the option to choose from different virtual reality setting depending on their preference (i.e., nature videos, meditations, interactive applications, among others).
  Interventions: Device: Virtual Reality; Other: Questionnaires
- Standard of care (Active Comparator): Participants will be asked to choose any activity of your preference during the chemotherapy session (i.e., watching tv, reading a book, listening to music or a podcast, etc.)
  Interventions: Other: Preferred activity; Other: Questionnaires

INTERVENTIONS:
Device: Virtual Reality — Virtual Reality Headset applied to the participants during chemotherapy session. Participants select their preferred virtual reality experience (i.e., nature videos, meditations, interactive applications, etc). Virtual reality (VR) by definition, is a simulated experience consisting of an experiential environment created by hardware and software technology capable of provoking sensations of real experiences. It can be further divided into 1) immersive; 2) semi-immersive; and 3) non-immersive. Immersive VR employs head-mounted display (HMD) system technology to separate users from their surroundings and engage in real-time with a three-dimensional environment generated by a computer.
  Arms: Virtual reality
Other: Preferred activity — Participants will engage in a preferred activity such as reading, watching television, coloring, etc. during chemotherapy.
  Arms: Standard of care
Other: Questionnaires — Participants will be administered multiple pre and post intervention questionnaires including NCCN Distress thermometer, GAD-7 and CCVA.

SUMMARY:
The goal of this clinical trial is to learn if the use of virtual reality during chemotherapy treatment helps participants achieve an improvement in distress, which may include unpleasant experience, anxiety, depression and/or pain.

Participants will:

* Be randomly assigned to one of two available groups (virtual reality or standard of care)
* Participations will only be during one chemotherapy session.
* Those assigned to virtual reality:

  * The research team will provide a virtual reality
  * The research team will provide guidance on how the headset works and will be available to assist with any questions or concerns.
  * Participants will also be able to choose different relaxing backgrounds depending on their preference. headset during the chemotherapy session for 15 to 30 minutes
* Those assigned to the standard of care:

  * The research team will provide the participants with the opportunity to choose a preferred activity such as reading a book, watching television, etc.

DETAILED DESCRIPTION:
In recent decades, new cancer cases have consistently risen. Participants diagnosed with cancer commonly face psychological symptoms including distress, anxiety, and depression in addition to physical symptoms (i.e., pain). Importantly, these symptoms might be exacerbated during chemotherapy sessions. New innovative technological strategies have been under development to control the symptoms and improve quality of life. Immersive virtual reality (VR) is a simulated experience that enables participants to interact with an artificial three-dimensional visual and auditory environment. VR could be an innovative intervention to relieve psychological symptoms associated with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Biopsy proven diagnosis of Cancer (any stage or type).
* Must have a National Comprehensive Cancer Network Distress Thermometer Score ≥ 5 any time since diagnosis.
* Must have the ability to understand and the willingness to sign a written informed consent document
* Followed by a medical oncologist, radiation oncologist, and/or breast surgeon at Cleveland Clinic.
* Ability to read and write in English or Spanish.

Exclusion Criteria:

* Age <18 years.
* No prior history of Cancer.
* Prior medical history of severe motion sickness.
* Prior medical history of seizures
* Pregnancy.
* Unable or unwilling to participate in the immersive Virtual Reality study at the Maroone Cancer Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in distress scores between pre- and post-intervention | Pre-intervention window of +/- 1 hours before intervention; post-intervention window of +/-1 hours post intervention
  The primary endpoint is the distress score change between pre- and post-intervention to evaluate the effectiveness of immersive virtual reality during chemotherapy sessions in reducing distress in participants with high levels of distress from baseline diagnosed with any type of Cancer, using The NCCN Distress Thermometer. This is a single-item questionnaire used to screen for psychological distress in participants. It consists of a simple scale ranging from 0 to 10, where participants rate their level of distress. A score of 5 or more on the NCCN Distress Thermometer indicates moderate to severe psychological distress

SECONDARY OUTCOMES:
Changes in pain scores between pre- and post-intervention | Pre-intervention window of +/- 1 hours before intervention; post-intervention window of +/-1 hours post intervention
  A secondary endpoint is the change in pain scores between pre- and post-intervention to evaluate the effectiveness of immersive virtual reality in reducing pain using the Universal Pain Assessment Tool. The Universal Pain Assessment Tool is a widely used instrument that consists of a visual analogue scale used to assess pain intensity. It includes a pain intensity scale that ranges from 0 to 10.
Changes in GAD-7 scores between pre- and post-intervention | Pre-intervention window of +/- 1 hours before intervention; post-intervention window of +/-1 hours post intervention
  A secondary endpoint is the change in anxiety scores pre- and post-intervention to evaluate the effectiveness of immersive virtual reality in reducing anxiety using the Generalized Anxiety Disorder-7 item (GAD-7). The Generalized Anxiety Disorder-7 item (GAD-7) questionnaires will be used to assess self-reported anxiety. The GAD-7 questionnaire will be interpreted as follows: minimal anxiety (0-4 points); mild anxiety (5-9 points); moderate anxiety (10-14 points) and severe anxiety (15-21 points).
Changes in CCVAS scores between pre- and post-intervention | Pre-intervention window of +/- 1 hours before intervention; post-intervention window of +/-1 hours post intervention
  A secondary endpoint is the change in depression scores pre- and post-intervention to evaluate the effectiveness of immersive virtual reality in reducing depression symptoms. The Cleveland Clinic Analog Scale (CCVAS) for depressive symptoms questionnaire will be used to assess self-reported depression. The CCVAS uses a 0-10 Likert scale, where 10 means feeling very depressed and 0 means not feeling any depression.
Predictor of intervention efficacy: Age | Day 1
  A secondary goal is to determine participants' clinical and sociodemographic characteristics associated with significant changes after the immersive virtual reality intervention. Age will be collected as a variable to assess whether this factor is a significant predictor of intervention efficacy.
Predictor of intervention efficacy: Race | Day 1
  A secondary goal is to determine participants' clinical and sociodemographic characteristics associated with significant changes after the immersive virtual reality intervention. Race will be collected as a variable to assess whether this factor is a significant predictor of intervention efficacy.
Predictor of intervention efficacy: Ethnicity | Day 1
  A secondary goal is to determine participants' clinical and sociodemographic characteristics associated with significant changes after the immersive virtual reality intervention. Ethnicity will be collected as a variable to assess whether this factor is a significant predictor of intervention efficacy.
Predictor of intervention efficacy: Martial Status | Day 1
  A secondary goal is to determine participants' clinical and sociodemographic characteristics associated with significant changes after the immersive virtual reality intervention. Marital status will be collected as a variable to assess whether this factor is a significant predictor of intervention efficacy.
Predictor of intervention efficacy: Occupation | Day 1
  A secondary goal is to determine participants' clinical and sociodemographic characteristics associated with significant changes after the immersive virtual reality intervention. Occupation will be collected as a variable to assess whether this factor is a significant predictor of intervention efficacy.
Predictor of intervention efficacy: Time since diagnosis | Day 1
  A secondary goal is to determine participants' clinical and sociodemographic characteristics associated with significant changes after the immersive virtual reality intervention. Time-to-diagnosis will be collected as a variable to assess whether this factor is a significant predictor of intervention efficacy.
Predictor of intervention efficacy: Current chemotherapy regimen | Day 1
  A secondary goal is to determine participants' clinical and sociodemographic characteristics associated with significant changes after the immersive virtual reality intervention. Participants' current chemotherapy regimen will be collected as a variable to assess whether this factor is a significant predictor of intervention efficacy.
Predictor of intervention efficacy: Time since therapy initiated | Day 1
  A secondary goal is to determine participants' clinical and sociodemographic characteristics associated with significant changes after the immersive virtual reality intervention. The "time since therapy was initiated" will be collected as a variable to assess whether this factor is a significant predictor of intervention efficacy.
Predictor of intervention efficacy: Attitudes towards use of virtual reality | Day 1
  A secondary goal is to determine participants' clinical and sociodemographic characteristics associated with significant changes after the immersive virtual reality intervention. Participant attitudes toward the use of virtual reality will be collected as a variable to assess whether this factor is a significant predictor of intervention efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Zeina Nahleh, MD FACP, Principal Investigator — Cleveland Clinic Florida, Maroone Cancer Center
Locations (1):
- Cleveland Clinic Florida, Maroone Cancer Center, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared as this is a minimally invasive pilot study.